CLINICAL TRIAL: NCT05973656
Title: Dissecting the Role of Acetaldehyde in Oral Carcinogenesis
Brief Title: Role of Acetaldehyde in the Development of Oral Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SPH-2021-29712; NCI-2022-09710 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2023-07-17; First posted 2023-08-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Alcohol-Related Carcinoma; Fanconi Anemia; Oral Cavity Carcinoma
MeSH Terms: conditions — Fanconi Anemia; Mouth Neoplasms | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (alcohol consumption) (Experimental): Participants who consume alcohol receive a standard drink or an alcohol dose that will result in a 0.03% BAC PO on study. Participants also undergo collection of saliva and breathalyzer testing throughout the trial.
  Interventions: Drug: Alcohol; Procedure: Biospecimen Collection; Procedure: Breath Test
- Group II (biospecimen collection) (Active Comparator): Participants who do not drink alcohol undergo collection of saliva, mouthwash, and cheek brush samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Breath Test

INTERVENTIONS:
Drug: Alcohol — Alcohol dose given orally that will result in a 0.03% blood alcohol concentration (BAC).
  Arms: Group I (alcohol consumption)
Procedure: Biospecimen Collection — Undergo saliva, mouthwash, and cheek brush collection
Procedure: Breath Test — Undergo breathalyzer testing

SUMMARY:
This is a minimal risk intervention study where healthy volunteers and individuals with Fanconi anemia will consume a single dose of alcohol and provide primarily non-invasive biological samples at various time points. Biospecimens to be collected include saliva, oral cells collected via mouthwash and cheek brush, and urine. The collection of two blood samples (5 mL each) will be optional and banked for future use.

ELIGIBILITY:
Inclusion Criteria:

* 21-45 years of age for alcohol drinkers
* Occasionally consume alcohol
* At least 1 drink per month for healthy volunteers
* At least 1 drink in the last 3 months for Fanconi anemia patients
* Meets one of the three criteria
* Healthy volunteer - ALDH2*1/1* homozygotes-not of Eastern Asian decent;
* Healthy volunteer - ALDH2*1/2* heterozygotes-of Eastern Asian decent and experience flushing when drinking
* Individual's with Fanconi anemia (FA).
* 18-45 years of age for non-drinkers
* Never consume alcohol/not had alcohol in the last 6 months
* Healthy volunteers.
* Non-smoker (smoked < 100 cigarettes in a lifetime)

Exclusion Criteria:

* Pregnant or nursing
* Taking any medication or drug that might affect alcohol use and absorption or that might be affected by alcohol consumption
* Healthy volunteers who have taken any antibiotics in the last 3 months
* Currently consuming more than 21 drinks per week
* Have any history of alcohol or drug related problems
* Current or former tobacco/nicotine product(s) user
* Any regular use of tobacco/nicotine products or marijuana in the last year (cigarettes, e-cigarettes, cigars, pipes, smokeless tobacco)
* "Trying" or limited use of any nicotine products or marijuana in the last 1 month
* Active infection (influenza, cold, COVID, respiratory / sinus infection) - admission in the study will be delayed pending improved health
* Non-FA volunteers who have an unstable medical condition or condition that could be affected by alcohol consumption (insulin-dependent diabetes, ulcers, heart issues)
* Experience severe adverse events (nausea, blacking out) when consuming even low doses of alcohol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Determine the acetaldehyde exposure to the oral cavity by comparing saliva levels before and after alcohol dose | Prior to alcohol dose, and 30 minutes, 1 hour, 2 hours, 4 hours, and 6 hours post alcohol dose
  Identify and quantify DNA adducts in the oral cells (mouthwash and cheek brush samples).

SECONDARY OUTCOMES:
Urine will be analyzed to confirm non-smoking status | Prior to alcohol exposure
  The optional blood samples will be analyzed for DNA adducts in the blood. We will measure the total concentration of the marker NNAL in urine.
Urine will be analyzed to confirm non-smoking status | Up to 6 hours after alcohol exposure
  The optional blood samples will be analyzed for DNA adducts in the blood. We will measure the total concentration of the marker NNAL in urine.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States